CLINICAL TRIAL: NCT03056716
Title: Silastic Versus Conventional Drain for Postoperative Drainage in Thoracic Surgery.
Brief Title: Silastic Versus Conventional Drain in Thoracic Surgery
Acronym: SD-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Serhat Yalcinkaya,MD, Assist. Prof. of Thoracic Surgery, T.C. Dumlupınar Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Silastic vs conventional drain
Record Dates: First submitted 2017-02-07; First posted 2017-02-17 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Air Leak From Lung; Post Procedural Persistent Drain Fluid
Keywords: thoracic surgery; silastic drains; conventional drains
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Silastic drain (Experimental): Placement of 19FR silastic drain as basal drain
  Interventions: Procedure: Silastic vs conventional drain in thoracic surgery
- Conventional drain (Active Comparator): Placement of 32FR conventional drain as basal drain
  Interventions: Procedure: Silastic vs conventional drain in thoracic surgery

INTERVENTIONS:
Procedure: Silastic vs conventional drain in thoracic surgery — Apical drains will be identical in size and material, and the basal drains will be different in groups. The patients will be followed for daily amounts of fluid drainage, duration of air leaks and fluid drainage, and duration of hospitalization, and the results will be compared statistically to asses any possible relationships with the outcome and the type of basal drain used.

SUMMARY:
In thoracic surgery, it is usual to place apical and basal drains for complete drainage of air and fluid out of the pleural cavity. The routinely used drains are mainly made of plastic. Recently silastic drains of smaller size are used without any complication. The investigators designed a prospective randomized trial to compare the draining properties of the two types of drains following various resections in thoracic surgery.

DETAILED DESCRIPTION:
Following the Institutional Review Board permission (permission no: 2009/27) the investigators started to recruit patients for the study in June 2009. Pneumonectomy, decortication, and diaphragm plication patients were not included in this study. The patients were consecutively placed in one of the two groups. In Group I, an apical 28FR size CD, and a basal 19FR SD were placed following surgery. In Group II, the apical drain was 28FR, and the basal drain was 32FR CDs. Basal drains were removed out when daily serous fluid drainage became 200 ml or less, and the apical were removed 48-72 hours following the cessation of air leak. The patients were discharged on the day after drain removal. The data concerning gender, age, diagnosis, operation side, type of operation, amount of fluid drainage, duration of fluid and air drainage, length of hospital stay, and complications if any, were noted.

ELIGIBILITY:
Inclusion Criteria:

* Candidates of surgery willing to participate in the experimental arm of the study and signing the informed consent form.

Exclusion Criteria:

* Pneumonectomy, diaphragm plication, and decortication candidates

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | 3 years
  Duration of hospital stay will be noted on the study datasheet and will be measured in days.

SECONDARY OUTCOMES:
Daily amount of fluid drainage | 3 years
  Daily amount of fluid drainage will be measured in mililiters during the daily rounds everyday, and will be noted on the datasheet.
Duration of fluid drainage | 3 years
  Everyday the drains will be checked for fluid drainage and the day without any drainage will be noted on the datasheet. Duration of fluid drainage will be measured in days since the postoperative day 1.
Duration of air leak | 3 years
  Everyday the drains will be checked for air leaks and the day without any air leak will be noted on the datasheet. Duration of air leak will be measured in days since the postoperative day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Research and Education Hospital, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient data except for the names and ID numbers will be shared.